CLINICAL TRIAL: NCT00004888
Title: A Safety and Efficacy Study of Doxil and Taxotere ± Herceptin in Advanced Breast Cancer
Brief Title: Combination Chemotherapy With or Without Trastuzumab in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02949; NCI-2012-02949 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E3198 (Other: Eastern Cooperative Oncology Group); E3198 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Results first posted 2011-11-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Docetaxel; Trastuzumab

ARMS (2):
- Arm I (combination chemotherapy) (Experimental): Patients receive doxorubicin hydrochloride liposome IV over 30 minutes followed by docetaxel IV over 1 hour. Treatment is repeated every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive maintenance therapy of docetaxel IV over 1 hour either weekly or every 3 weeks. Maintenance continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Drug: docetaxel; Other: laboratory biomarker analysis
- Arm II (combination chemotherapy, trastuzumab) (Experimental): Patients receive trastuzumab IV over 90 minutes on day 1, with subsequent doses over 30 minutes. Patients receive doxorubicin HCl liposome IV over 30 minutes followed by docetaxel IV over 1 hour on day 2 of course 1, followed by subsequent doses on day 1 of each course. Antibody therapy continues weekly and chemotherapy every 3 weeks for 8 courses.
  Patients may receive maintenance therapy of trastuzumab IV over 30 minutes weekly followed by docetaxel IV over 1 hour weekly or every 3 weeks. Maintenance continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Drug: docetaxel; Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
  Arms: Arm II (combination chemotherapy, trastuzumab)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combination chemotherapy with or without trastuzumab in treating women who have metastatic breast cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and feasibility of the combination of liposomal doxorubicin (Doxil) and Taxotere (Taxotere) ± trastuzumab (Herceptin), particularly with respect to cardiotoxicity.

II. To evaluate the overall objective response rate, response duration, time to treatment failure, and median survival of patients with metastatic breast cancer treated with Doxil and Taxotere ± Herceptin.

III. To determine the overall toxicity of Doxil and Taxotere ± Herceptin in patients with advanced breast cancer.

IV. To determine whether there is an association between trough plasma levels of cTnT (cardiac troponin T) and NT-proBNP (brain natriuretic peptide) and any cardiac event (CHF or LVEF decrease).

V. To determine tissue and plasma levels of HER2 using several assays and explore potential correlation with protocol treatment toxicity and/or response.

OUTLINE: Patients are assigned to one of two treatment arms according to HER2 overexpression status.

Arm I (HER2 nonoverexpressed): Patients receive doxorubicin hydrochloride liposome IV over 30 minutes followed by docetaxel IV over 1 hour. Treatment is repeated every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.

Patients may receive maintenance therapy of docetaxel IV over 1 hour either weekly or every 3 weeks. Maintenance continues in the absence of disease progression or unacceptable toxicity.

Arm II (HER2 overexpressed): Patients receive trastuzumab IV over 90 minutes on day 1, with subsequent doses over 30 minutes. Patients receive doxorubicin HCl liposome IV over 30 minutes followed by docetaxel IV over 1 hour on day 2 of course 1, followed by subsequent doses on day 1 of each course. Antibody therapy continues weekly and chemotherapy every 3 weeks for 8 courses.

Patients may receive maintenance therapy of trastuzumab IV over 30 minutes weekly followed by docetaxel IV over 1 hour weekly or every 3 weeks. Maintenance continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 89 patients were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast with manifestations of metastatic progression
* HER2 expression status in primary breast tissue and/or site(s) of metastasis must be determined by the ECOG Pathology Coordinating Office; (these are the results that will be used at time of registration); NOTE: for this protocol, HER2/neu non-overexpressed status will be defined as 0 and 1+ scores using the DAKO HercepTest; HER2 overexpressed status will be defined as 2+ score (if confirmed amplified by FISH) or 3+ score using the DAKO HercepTest
* Cytologically positive pleural or peritoneal effusions are considered evaluable disease provided local intra-cavitary treatment is not introduced at the onset of therapy; to be considered as evaluable disease, pleural effusions may not have been previously drained or sclerosed
* Blastic or mixed blastic/lytic osseous metastases only are evaluable disease provided they are accompanied by an analgesic requirement or a decrease in performance status, and will not require radiation treatment within two cycles from the start of protocol; pure osteolytic disease is evaluable; bone disease must be x-ray proven for the site to be evaluable; patients whose only evidence of metastatic disease is an abnormal bone scan without confirmatory x-rays are not eligible for this study
* No prior chemotherapy for advanced disease; prior adjuvant chemotherapy (including taxanes) allowed, if completed > 6 months before the diagnosis of metastatic disease; no prior adjuvant anthracycline, nor any prior exposure to other anthracycline- (e.g., epirubicin, any liposomal doxorubicin formulation), nor any anthracenedione- (e.g., mitoxantrone) containing regimen allowed; no prior therapy with Herceptin allowed; NOTE: chemotherapy after ipsilateral breast recurrence following breast conservation surgery would not be considered chemotherapy for advanced disease; however, in post-mastectomy patients chemotherapy for local/regional recurrence is considered treatment for advanced disease
* No prior radiotherapy other than to the conserved breast, to the post-mastectomy chest wall, or to a limited field involving < 25% of marrow-containing bone; NOTE: previous post-mastectomy radiation therapy involving chest wall ± internal mammary lymph node chain (IMN) is allowed; however, patients who received photon IMN treatment are ineligible; NOTE: radiotherapy must be completed >= 2 weeks prior to registration; it may not be given concurrently with Doxil, Taxotere, or Herceptin
* Prior hormonal therapy in either a metastatic or adjuvant setting is allowed, but patients must have been off such therapy for >= 2 weeks prior to registration
* Disease-free of prior non-breast invasive malignancies for >= 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* ECOG performance status of 0, 1, or 2
* At least two weeks after any major surgery (including mastectomy) and recovered from all toxicity
* Creatinine =< 1.5 mg/dl
* Granulocytes >= 1,500/mm³
* Platelets >= 100,000/mm³
* SGOT(AST) =< 2.5 x the upper limit of normal
* Bilirubin within normal limits for institution
* No history of deep venous thrombosis, pulmonary thromboembolism, or other thromboembolic condition
* Women must not be pregnant or breastfeeding; the effect of Herceptin to the fetus is unknown; Doxil is known to be harmful to the fetus
* Women of childbearing potential must be advised to use an accepted and effective method of contraception
* No patients with untreated brain metastasis or brain metastasis undergoing radiation or for whom brain metastasis represent the sole site of disease; patients with previously treated brain metastasis who have responded to brain radiotherapy and/or surgery and continue in response are eligible, provided the brain is not the only site of disease
* The left ventricular ejection fraction must be at or above the lower institutional limits of normal (as assessed by MUGA scan or echocardiogram obtained within six weeks prior to registration); patient will not be eligible if baseline LVEF assessment not performed
* No prior history of myocardial infarction, congestive heart failure, or arrhythmia requiring medication; no history of hypertension or systolic or diastolic dysfunction; no EKG evidence of ventricular hypertrophy, conduction abnormality, or serious arrhythmia; patient will not be eligible if baseline EKG assessment not performed within 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-01; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Wolff, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on Oct 19, 2000 and closed on Sept 7, 2004. Accrual to Arm II was suspended on April 23, 2002 for a pre-planned interim analysis regarding cardiac safety and resumed on Nov 6, 2002. Study participants all came from ECOG institutions.
Pre-assignment Details: Entry on the study requires determination by the Eastern Cooperative Group Pathology Coordinating Office of HER2 expression status in primary breast tissue or site of metastasis. Patients with PS 2 were excluded from further enrollment in both arms as they were found to experience more severe toxicities and more frequent dose reductions.
Groups:
- Arm I: Doxorubicin and Taxotere: Patients received PLD 30 mg/m^2 IV followed by docetaxel 60 mg/m^2 IV, one hour after PLD completion, every 3 weeks for a total of 8 cycles. Dexamthasone 8 mg orally twice a day was administered the day before, the day of, and the day following docetaxel. The maximum allowed cumulative dose of PLD was 240 mg/m^2. Pyridoxine 200 mg PO daily started on Day 1 of Cycle 1 and continued daily while the patient was on PLD.
- Arm II: Doxorubicin, Taxotere, and Herceptin: Patients received the weekly antibody therapy with trastuzumab in addition to the induction chemotherapy with PLD and docetaxel every 3 weeks as outlined for Arm I above for a total of 8 cycles. Trastuzumab was administered 4 mg/kg IV on Day 1, then 2 mg/kg IV weekly.
Period: Overall Study
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Started | 38 (Of the 41 pts, 3 were ineligible.) | 46 (Of the 48 pts, 2 were ineligible.)
Completed | 27 | 22
Not Completed | 11 | 24
Not completed — Adverse Event | 5 | 10
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Progressive Disease | 4 | 9
Not completed — Death without progressive disease | 0 | 1
Not completed — Toxic death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin | Total
Number analyzed (Participants) | 38 | 46 | 84
Age, Continuous [Median (Full Range); unit: years] | 53 [33 to 80] | 53 [23 to 80] | 53 [23 to 80]
Sex/Gender, Customized [Number; unit: participants] — All participants are female.
  participants
    Female | 38 | 46 | 84

OUTCOME MEASURES:

1. Primary Outcome: Grades of Cardiotoxicity Events in the Subset of Patients Reporting a Cardiotoxicity Event
Description: This table summarizes the cardiotoxicity events of different grades. Grade 1 is a decline of left ventricular ejection fraction(LVEF) >=10% but <20% of baseline value. Grade 2 is LVEF below LLN (50%) or decline of LVEF >=20% of baseline value. Grade 3 is congestive heart failure responsive to treatment. Please note that only a subset of patients reported cardiotoxic events so the totals will not add up to the total number of participants.
Time Frame: Baseline, after cycle 4 (~84 days), after cycle 8 (~168 days), and 30 or more days after last cycle of induction therapy
Population: Treated patients who had a cardiotoxicity event
Measure: Number; unit: participants
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Number analyzed (Participants) | 16 | 37
participants
  Grade 1 After Cycle 4 (approx. 84 days) | 2 | 12
  Grade 1 After Cycle 8 (approx. 168 days) | 4 | 8
  Grade 1 After 30 days or more after last cycle | 1 | 10
  Grade 2 After Cycle 4 (approx 84 days) | 3 | 0
  Grade 2 After Cycle 8 (approx 168 days) | 4 | 2
  Grade 2 After 30 days or more after last cycle | 1 | 5
  Grade 3 After Cycle 4 (approx 84 days) | 1 | 0
  Grade 3 After Cycle 8 (approx 168 days) | 0 | 0
  Grade 3 After 30 days or more after last cycle | 0 | 0

2. Secondary Outcome: Best Overall Response Using Eastern Cooperative Group Solid Tumor Response Criteria.
Description: Please note that overall response includes CR and PR. CR is defined as complete disappearance of all clinically detectable malignant disease for at least 4 weeks. PR is greater than or equal to 50% decrease in tumor size for at least 4 weeks without increase in size of any area of known malignant disease of greater than 25%, or appearance of new areas of malignant disease. No change is defined as no significant change in measurable or evaluable disease for at least 4 weeks. Progression is defined as a significant increase in size of lesions present at the start of therapy or after a response.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually until death or until reaching full study stop date. Data as of Nov 21, 2007 is used for this report. Please note that best overall response is reported in the table.
Population: Eligible Patients
Measure: Number; unit: participants
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Number analyzed (Participants) | 38 | 46
participants
  Complete Response | 1 | 4
  Partial Response | 17 | 17
  No Change | 11 | 11
  Progression | 6 | 9
  Unevaluable | 3 | 5
Statistical Analysis 1: Comparison: Arm I: Doxorubicin and Taxotere; Test type: Superiority or Other; Overall Response Rate = 0.474, 95% CI 2-sided [0.31 to 0.642]
Statistical Analysis 2: Comparison: Arm II: Doxorubicin, Taxotere, and Herceptin; Test type: Superiority or Other; Overall Response Rate = 0.457, 95% CI 2-sided [0.309 to 0.61]

3. Secondary Outcome: Overall Survival
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually until death or until reaching full study stop date. Data as of November 21, 2007 is used for this report.
Population: All eligible patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Number analyzed (Participants) | 38 | 46
months | 24.6 [14.7 to 37.3] | 31.8 [23.7 to 44.9]

4. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival was defined as time from study entry to progression or to death without documentation of progression. A progression is defined as a significant increase in size of lesions present at the start of therapy or after a response.
Time Frame: as for outcome 3
Population: All eligible patients were included in this analysis. Please note that 2 patients on Arm B died without documentation of progression. Also, 4 patients died or were taken off treatment before follow-up evaluations, and PFS was censored at zero.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Number analyzed (Participants) | 38 | 46
months | 11 [8.6 to 12.8] | 10.6 [5.6 to 15.7]

5. Primary Outcome: Summary of Left Ventricular Ejection Fraction Values
Description: This table summarizes the LVEF information at baseline, post Cycle 4, post Cycle 8, and 30 or more days after Cycle 8 on all treated patients and on the eligible subset. LVEF drops reported are absolute (not relative) drops.
Time Frame: Baseline, after cycle 4, after cycle 8, and 30 or more days after last cycle of induction therapy.
Population: All treated patients
Measure: Mean (Standard Deviation); unit: LVEF percent
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Number analyzed (Participants) | 41 | 48
LVEF percent
  Baseline | 64.8 (8.3) | 62.9 (7.2)
  Post Cycle 4 | 63 (7.9) | 61.7 (7.2)
  Post Cycle 8 | 60.8 (8.2) | 58.9 (7.4)
  greater than or equal to 30 days after cycle 8 | 62.6 (6.4) | 59.1 (7.5)
  Baseline minus post cycle 4 | 2.3 (7.5) | 1.6 (8.0)
  Baseline minus post cycle 8 | 4.2 (8.8) | 4.9 (6.7)
  Baseline minus 30 days or more after cycle 8 | 0.9 (7.1) | 6.2 (9.4)

6. Secondary Outcome: Duration of Response
Description: Defined as time from onset of PR or CR, whichever occurred first, until objective evidence of progression.
Time Frame: as for outcome 3
Population: Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Number analyzed (Participants) | 18 | 21
Months | 10.1 [6.7 to 15.4] | 14.7 [7.8 to 23.7]

ADVERSE EVENTS:
Time Frame: Information about toxicities was collected during treatment for all treated patients and the table shows toxicities experienced by patients. These are limited to toxicities reported on case report forms. The average time period was 5-6 months.
Description: Please note that all of these toxicities are considered at least possibly treatment related by the study chair.
Arm/Group | Arm I: Doxorubicin and Taxotere | Arm II: Doxorubicin, Taxotere, and Herceptin
Serious Adverse Events (participants affected / at risk) | 41/41 | 48/48
Other Adverse Events (participants affected / at risk) | 41/41 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Doxorubicin and Taxotere (N=41) | Arm II: Doxorubicin, Taxotere, and Herceptin (N=48)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 9 (9) | 18 (26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 22 (83) | 28 (82)
Neutropenia (Blood and lymphatic system disorders) | 24 (88) | 32 (120)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular Arrhythmias (Cardiac disorders) | 1 (1) | 0 (0)
Infection with Grade 3 or 4 neutropenia (Infections and infestations) | 5 (5) | 6 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (8) | 6 (10)
Thrombosis/embolism (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infection with Unknown ANC (Infections and infestations) | 3 (3) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (9) | 8 (9)
DIC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Stomatitis (General disorders) | 7 (7) | 11 (13)
Diarrhea without prior colostomy (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bilirubin Increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
AST Increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Tearing (Eye disorders) | 2 (2) | 0 (0)
abdominal pain (General disorders) | 1 (1) | 0 (0)
Creatinine Increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Doxorubicin and Taxotere (N=41) | Arm II: Doxorubicin, Taxotere, and Herceptin (N=48)
Allergic Reaction (General disorders) | 3 (3) | 8 (11)
Anemia (Blood and lymphatic system disorders) | 30 (331) | 39 (586)
Leukopenia (Blood and lymphatic system disorders) | 31 (204) | 43 (267)
Neutropenia (Blood and lymphatic system disorders) | 22 (72) | 36 (109)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (56) | 6 (22)
Cardiac-left ventric (Cardiac disorders) | 9 (10) | 11 (15)
Edema (Skin and subcutaneous tissue disorders) | 6 (13) | 5 (15)
Fatigue (General disorders) | 29 (128) | 33 (68)
Fever (General disorders) | 5 (7) | 6 (8)
Rigors/Chills (General disorders) | 5 (8) | 6 (10)
Weight Loss (General disorders) | 3 (6) | 8 (11)
Alopecia (General disorders) | 31 (225) | 38 (220)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 20 (58) | 30 (96)
Nail Changes (General disorders) | 17 (51) | 18 (80)
Pigmentation (General disorders) | 4 (16) | 5 (11)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (13) | 10 (18)
Hot Flashes (General disorders) | 2 (4) | 9 (23)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 11 (22)
Constipation (Gastrointestinal disorders) | 9 (13) | 16 (37)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 7 (26)
Nausea (General disorders) | 22 (53) | 31 (104)
Stomatitis (General disorders) | 28 (98) | 38 (108)
Taste Disturbance (General disorders) | 6 (53) | 6 (21)
Vomiting (Gastrointestinal disorders) | 11 (16) | 18 (33)
Diarrhea (Gastrointestinal disorders) | 13 (20) | 21 (42)
Bilirubin Increased (Hepatobiliary disorders) | 2 (4) | 2 (3)
Hypoalbuminemia (Hepatobiliary disorders) | 2 (5) | 1 (1)
AST Increased (Blood and lymphatic system disorders) | 21 (60) | 24 (59)
Infection with neutro (Infections and infestations) | 3 (6) | 11 (22)
Dizziness/lightheaded (General disorders) | 8 (9) | 2 (3)
Insomnia (General disorders) | 4 (13) | 4 (8)
Neuropathy Sensory (Nervous system disorders) | 16 (33) | 17 (39)
Conjunctivitis (Eye disorders) | 3 (5) | 1 (1)
Dry Eye (Eye disorders) | 4 (4) | 2 (12)
Tearing (Eye disorders) | 15 (46) | 15 (41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (22) | 8 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (31) | 12 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less